CLINICAL TRIAL: NCT05885542
Title: Sex Differences in the Interface Between Cannabis Use and Stress Among Emerging Adults
Brief Title: SCORE Emerging Adult Cannabis Use & Stress
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kevin Gray, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00127995
Record Dates: First submitted 2023-04-03; First posted 2023-06-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Cannabis Use Disorder
Keywords: cannabis; stress; sex; withdrawal
MeSH Terms: conditions — Marijuana Abuse; Coitus | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either double-blind single-dose CBD 800 mg or matched placebo (1:1) utilizing a stratified random block design. Randomization will be stratified by biological sex (female, male) to facilitate analyses incorporating sex as a biological variable.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization allocation will be completed by statisticians in the Biostatistics Resource Core and all other investigators, study personnel, and participants will be blinded to past and future study allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- cannabidiol 800 mg (Experimental): Cannabidiol 800 mg will be administered orally once in the laboratory prior to a stress induction paradigm.
  Interventions: Drug: Cannabidiol oral solution
- placebo (Placebo Comparator): Placebo (formulated to appear identical to active condition) administered orally once in the laboratory prior to a stress induction paradigm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol oral solution — Double-blind cannabidiol oral solution 800 mg administered once
  Arms: cannabidiol 800 mg
Drug: Placebo — Double-blind placebo oral solution administered once
  Arms: placebo

SUMMARY:
The interface between cannabis use and stress is a particularly important focus for sex differences research in emerging adults. Given the dynamics at play in this critical stage when cannabis use is most prevalent, developmentally informed research is needed to guide tailored clinical interventions. This study will apply rigorous and innovative methods to elucidate sex differences in the nexus of cannabis use and stress among emerging adults with cannabis use disorder to guide the development of tailored treatments.

DETAILED DESCRIPTION:
Among the physiological systems most important to brain development in emerging adulthood is the endocannabinoid system, which among other roles facilitates cognitive and behavioral processing, including the underpinnings of stress management and resiliency. Sex differences in endocannabinoid system development have been identified, and emerging evidence indicates a bidirectional relationship between stress exposure and the endocannabinoid system during emerging adulthood. Repeated exposure to exogenous cannabinoids, such as those administered via cannabis use, perturbates endocannabinoid system development, which may adversely affect the programming of future coping in a manner that differs by sex. Use of cannabis, which exerts its psychoactive effects via delta-9-tetrahydrocannabinol binding to endocannabinoid receptors, is more common among emerging adults than in any other age group. Many regular users develop a maladaptive, impairing pattern of use characterized as cannabis use disorder (CUD). A constellation of preliminary evidence suggests several factors disproportionately complicate CUD in females compared to males; the salience of these factors in emerging adulthood indicates that this developmental stage deserves focused sex differences research to inform clinical management. A central running thread is the importance of stress and stress-reactivity across endocannabinoid system development, cannabis use, CUD, cannabis withdrawal, and relapse to cannabis use. This study combines rigorous ecological momentary assessment (EMA), controlled human laboratory procedures, and innovative bioassay collection. Emerging adult cannabis users with CUD (ages 18-25, N=148, 1:1 female to male ratio) will undergo 3 days of reinforced abstinence with EMA monitoring of cannabis withdrawal and stress-related symptoms, followed by a standardized laboratory stress induction paradigm. Blood levels of endocannabinoid system markers will be assessed before and after the abstinence period; during the lab session, self-report measures and biomarkers of stress reactivity will be collected. Double-blind cannabidiol (CBD) versus placebo dosing before the laboratory stress paradigm will allow for examination of effects on stress response during withdrawal. Prior work indicates CBD administration reduces stress response in general populations and preliminary research suggests this effect may extend to cannabis users; this has not been rigorously applied to induced stress amid cannabis withdrawal in emerging adults with CUD, a context particularly important for females with CUD who often report using cannabis to cope with stress. Following the laboratory session, EMA monitoring will resume as participants return to ad libitum cannabis use, providing the opportunity to test associations between stress reactivity and time to resumption of use. The proposed study is designed to elucidate sex differences and guide the development of tailored treatments that address factors disproportionately affecting emerging adult females with CUD.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments
* Meet DSM-5 criteria for CUD and report using cannabis at least five times weekly over the past month. While individuals may also meet criteria for other mild substance use disorders, they must identify cannabis as their primary substance
* Age 18-25
* BMI between 18-30 (to decrease variability in CBD response and in endocannabinoid system measures)
* AST, ALT, and total bilirubin within the laboratory reference range of normal
* Consent to alcohol abstinence for 12 hours prior to study visits, three days of cannabis abstinence as part of study procedures, and abstinence from all substances aside from cannabis, alcohol, and nicotine for the duration of the study
* Sexually active females of childbearing potential must agree to utilize an effective means of birth control.
* Consent to random assignment to CBD versus placebo

Exclusion Criteria:

* Females who are pregnant, nursing, or planning to become pregnant during the study.
* Current severe substance use disorder other than cannabis
* Current medications or supplements with clinically significant interactions with cannabidiol (per Lexicomp, this list includes Blasting, Doxorubicin, Mavacamten, Pazopanib, Sirolimus, Topotecan, Vincristine, Afatinib, Berotraslstat, Cilostazol, Citalopram, Colchicine, Digoxin, Lefamulin, Relugolix, Relugolix+Estradiol+Norethindrone, Rimegepant, Tizanidine, Ubrogepant, and Venetoclax in the categories of "avoid combination" or "consider therapy modification")
* Current unstable psychiatric or medical disorder that would interfere with safety, compromise data integrity, or preclude reliable participation
* History of hypersensitivity to CBD, sesame, or sesame products
* Inability to comply with study procedures

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All
Enrollment: 148 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Cannabis withdrawal symptoms | Assessed after 3-day cannabis abstinence period
  Cannabis Withdrawal Scale score (Allsop et al., 2011) [minimum score 0 and maximum score 190; higher score means a worse outcome]
Stress reactivity | Measured 5 minutes after laboratory-administered Trier Social Stress Task
  Within Session Rating Scale - Stress score (Childress et al., 1986) [minimum score 0 and maximum score 10; higher score means a worse outcome]
Time to resumption of cannabis use | Measured as the time span from laboratory session to time of resumption of ad lib cannabis use (maximum of 10 days)
  After 3-day abstinence phase and laboratory session, ecological momentary assessment will be conducted twice daily for a 10-day span. Participants may resume ad lib cannabis use, and will be prompted to self-report the day/time that they resume cannabis use [minimum score 0 and maximum score 10 days, with the possibility of no resumption at all; higher score means a better outcome, and no resumption at all by the end of the 10 days is the best possible outcome]

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Gray, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
A final de-identified data set will be made available for retrieval and analysis.